CLINICAL TRIAL: NCT00633503
Title: Monitoring of Tissue Transfer Flaps by Modulated Imaging (MI) Spectroscopy
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Responsible Party: Principal Investigator, Gregory R. Evans, Professor, University of California, Irvine
Other Study IDs: 2007-5891
Record Dates: First submitted 2008-03-04; First posted 2008-03-12 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-04

CONDITIONS: Reconstructive Surgical Procedures; Tissue Transplantation
Keywords: free tissue transfer; pedicle tissue transfer; complications; modulated imaging spectroscopy; observation; clinical observation/diagnosis; tissue defects requiring free tissue transfer; tissue defects requiring pedicle tissue transfer
MeSH Terms: conditions — Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A-Observation: All patients undergoing pedicle and free tissue transfer.

SUMMARY:
Tissue transfer flaps are a method of moving tissue from a donor location to a recipient location. In the case of a free tissue transfer flaps, the blood vessels to the transferred tissues are detached and then re-attached to different arteries & veins at the recipient site. The process of reconstructive surgery using tissue transfer flaps allows for improved results in terms of functionality, aesthetic appearance, and psychological well-being in patients requiring reconstructive surgery after cancer resection or trauma. The process of reconstructive surgery using tissue transfer flaps is not without complications. These complications may include acute arterial or venous occlusion, as well as the development of late complications such as fat necrosis and flap atrophy.

The purpose of this pilot study is to determine if a novel, unique, portable, non-contact optical imaging device developed at the Beckman Laser Institute called Modulated Imaging (MI) can detect changes in a flap's optical properties, which can correlate with arterial or venous occlusion or with the development of fat necrosis or flap atrophy. The study would also evaluate if changes in the tissue transfer flap's optical properties, as detected by the device could be employed as a monitoring device in the post-operative period after reconstructive surgery. The MI device's detection of specific optical properties of a tissue flap could also potentially be used as a diagnostic tool to predict the likelihood of the development of fat necrosis or flap atrophy in a delayed fashion several months after reconstructive surgery.

Prior animal and clinical studies using similar devices have demonstrated that changes in the total hemoglobin concentration and percentage of oxygenated hemoglobin in the tissue transfer flap can be used to differentiate between arterial and venous occlusion. These other similar devices have been shown to be able to detect venous occlusion prior to clinical manifestations of venous occlusion using standard monitoring methods. This early detection of venous occlusion has important implications. It is well established that early detection and surgical re-exploration and correction of venous occlusion is associated with improved survival and salvage rates of tissue transfer flaps. It has been suggested in the reconstructive literature that the development of fat necrosis and flap atrophy are caused by a relative arterial or venous insufficiency, which could be detected using the MI device prior to the clinical manifestations of these complications.Patients undergoing reconstructive surgery at UCI Medical Center will be recruited for enrollment into the study. The study design requires following the patients and review their medical records in order to determine the clinical outcomes of their reconstructive surgery. The process of review of the medical record will require the review of both the in-patient medical record during the hospitalization in which the reconstructive surgery takes place and the outpatient medical record after surgery in order to observe for the possible development of the acute and delayed complications of reconstructive surgery.

DETAILED DESCRIPTION:
Objectives:

1. To develop a safe, non-contact, intra-operative & post-operative device, which can be used as an adjunct to the clinical evaluation of tissue transfer flaps after reconstructive surgery.
2. To develop an adjunctive device that can reliably detect and distinguish arterial and venous occlusion before the clinical manifestations of such occlusions, and thus provide the scientific basis for future studies which may use the device to potentially improve the salvage rates after re-exploration for such complications.
3. To evaluate if changes in the optical properties of tissue transfer flaps during the immediate post-operative period can be used to predict the development of late complications of tissue transfer flaps, such as the development of fat necrosis and/or flap atrophy.

Specific aims:

1. To record intra-operative and post-operative images of pedicle and free tissue transfer flaps used in reconstructive surgery with a device that shines low energy near infrared light that is spatially modulated into a sinusoidal configuration of amplitude called Modulated Imaging (MI).
2. To study if the MI device described above is able to collect data regarding the optical properties of the tissue transfer flaps, which can then be used to detect acute post-operative occlusion of the artery or of the vein going to and from the tissue transfer flap.
3. To study if there is a correlation between the immediate post-operative optical properties of tissue transfer flaps and the development of late complications such as fat necrosis and flap atrophy.

Hypotheses:

1. Prior authors have demonstrated that tissue spectroscopy can be used in both animal & human experiments to detect and differentiate between tissue transfer flaps with adequate vascular supply vs. flaps with either artery and/or vein occlusions prior to the detection of such complications using standard clinical observation during the post-operative period. These authors demonstrated that detection of the changes from baseline values in the post-operative period of the total hemoglobin [Hb-total], deoxygenated hemoglobin [Hb-deoxy], and oxygenated hemoglobin [Hb-O2] concentrations using tissue spectroscopy correlated with the clinical development of arterial or venous occlusion. 1,2 As the MI device developed at the Beckman Laser Institute has been demonstrated to be able to detect the [Hb-total], [Hb-deoxy] and [Hb-O2] as well as the concentration of water,[H2O] in a non-contact manner; we believe the MI device will also be able to detect development of arterial and/ or venous occlusion in tissue transfer flaps without requiring direct tissue contact with a tissue spectroscopy device, as was the case with the instruments used by other authors.3, 4
2. There are higher rates of fat necrosis and flap atrophy that occur after specific types of free tissue transfer flaps, [i.e., higher rates occur with Deep Inferior Epigastric Perforator (DIEP) flaps vs. Transverse Rectus Abdominis (TRAM) flaps.5, 6 Some authors have suggested that early flap congestion and the development of late fat necrosis may be due to venous insufficiency, without complete venous occlusion 7. We hypothesize that early post-operative changes in the flap's optical properties may be used to predict the development of late complications such as fat necrosis and flap atrophy, as these complications are thought to be due to a relative arterial and/or venous insufficiency to the tissue transfer flap; and thus should be reflected in the tissue's optical properties as detected by the MI device.

Rationale: The use of tissue pedicle and free tissue transfer flaps allows for increased reconstructive possibilities for patients that have had disfigurement or loss of function after trauma or oncological surgical resection. Generally, the process of creating a pedicle tissue transfer flap involves the isolation of tissues onto a single artery and vein and then rotating this tissue from the donor site to the site requiring reconstruction. A free tissue transfer flap involves a process similar to the creation of a pedicle flap except that the artery and vein going to the flap's tissues are divided and re-implanted at the site of reconstruction. This process of using tissue transfer flaps however has known complications, including acute complications such as arterial or venous occlusion and late complications such as the development of fat necrosis and flap atrophy.

Acute complications involving the vascular structures of the flap can be either partial or complete occlusion of the artery or vein going to and from the tissue flap. Both pedicle and free tissue transfer flaps can develop severe complications if either the artery or vein is compromised, including complete death of the tissue in the flap. If the vascular structures going to the flap(s) are compromised then the tissues used for reconstructive surgery may undergo damage. This tissue damage can become extensive and result in the loss of part or the entire tissue mass in the tissue transfer flap, which in turn can result in increased morbidity and mortality to the patient. In the reconstructive surgery literature, it has been shown that frequent monitoring during the first 48-72 hours after reconstructive surgery allows for early detection and intervention when a vascular compromised flap occurs. This earlier detection then can translate into earlier interventions including surgical re-exploration, which has been shown to improve the salvage rates of vascular compromise of the tissue transfer flaps.8, 9 It is generally known that venous thrombosis has a worse out-come, when compared to arterial thrombosis after surgical re-exploration and reestablishment of blood flow. This difference between arterial and venous thrombosis is thought to be due to the differences in the pathophysiology involved in venous congestion. In venous thrombosis tissue fluid content is increased due to initially continued arterial inflow, thus when venous out-flow is re-established the tissue edema continues to inhibit the diffusion of oxygen through the interstitial space from the capillaries to the tissue cells in the vascular beds were edema remains. The fact that venous thrombosis is more difficult to clinically detect early may also contribute to the poorer prognosis associated with venous thrombosis when compared to arterial thrombosis.10

Given the difficulty of early detection of venous thrombosis, and of the decreased rates of successful salvage after surgical re-exploration for venous thrombosis, authors have employed successfully the use of tissue spectroscopy to detect venous thrombosis several hours before the clinical manifestations of thrombosis 2. These authors employed a spectroscopy device, which requires direct contact with the tissues being evaluated and only provided a small surface area in which the tissue flap's optical properties were measured. The device, however, is able to provide both diffuse optical tomography and rapid wide-field quantitative mapping of the tissue's optical properties in a single measurement platform through a device that does not require direct contact with the tissues being evaluated 3, 11. As theMI device is a new novel device developed at the Beckman laser Institute and has not been used to evaluate human tissue transfer flaps this would be a pilot study. This pilot study would seek to determine if this specific device is also able to detect vascular occlusion prior to clinical detection of such occlusion, as well as to differentiate between arterial and venous occlusions in a similar manner to other devices used by other authors, which employed tissue spectroscopy to monitor tissue transfer flaps.

As mentioned above, delayed complications can develop after tissue transfer flaps are used in reconstructive surgery, which include fat necrosis and flap atrophy. These late complications are thought to be caused by a relative vascular insufficiency supplying the flaps. It is proposed that the increased venous congestion and increased rates of fat necrosis with the use of DIEP flaps when compared to TRAM flaps in breast reconstruction is due to a relative venous insufficiency that is not diminished enough to cause flap loss, but is on occasion great enough to result in the development of fat necrosis 7. The late development of flap atrophy may also be due to a relative arterial or venous insufficiency that occurs at the time of surgical reconstruction, and results in a relative global tissue flap ischemia leading to the development of flap atrophy. One of the goals of this experiment is to determine if any characteristic of the optical properties in a tissue transfer flap in the near post-operative setting can predict the development of either fat necrosis or flap atrophy.

The MI device is a novel unique device when compared to other spectroscopic devices used to study tissue transfer flaps. MI uses a non-contact optical imaging technology developed at the Beckman Laser Institute that has the unique capability of performing both diffuse optical tomography and rapid, wide-field quantitative mapping of tissue optical properties within a single measurement platform. While other non-contact spectroscopic devices use a time-modulation methods, MI alternatively uses spatially modulated illumination for imaging of tissue constituents. The MI system consists of 1) a light projection system that illuminates the tissue with spatial sinusoid patterns, and 2) a CCD camera, which collects the diffusely reflected light in a non-contact geometry. The wavelength of illumination can be selected by bandpass filtering of a broadband source (i.e. tungsten lamp), or by use of a monochromatic source (i.e. laser diode). Lastly, tissue fluorescence measurements can be performed by placing a combination of source-blocking and bandpass emission filters in front of the camera. 3, 11

The diffusely reflected amplitude of the modulated wave carries both optical property (absorption, fluorescence, scattering) and depth information. Specifically, the sampling depth of the spatially modulated wave is a function of the frequency of illumination and the tissue optical properties. This shares many analogies to the broadband frequency-domain photon migration (FDPM) approach. {12, 13} Consequently, measurement of multiple spatial frequencies (periodicities) allows MI to perform two functions. First, use of a wide range of frequency patterns allows depth-selective imaging and thus tomography of the internal 3D tissue structure. Secondly, it can rapidly and quantitatively map optical absorption, fluorescence yield, and scattering coefficients in near-real time, with high resolution and over a wide field-of-view.

The ability to separate optical absorption from scattering distinguishes MI from conventional planar reflectance imaging methods. Absorption and scattering maps can be used to characterize the tissue's biochemical composition and structure. We have shown that these intrinsic tissue contrast elements vary with tissue types, and their wavelength dependence provides spectral "fingerprinting" that can be used to delineate the spatial relationships among tissues with different optical properties and can be used to determine the amount of H2O, [Hb-total], [Hb-deoxy], [Hb-O2] & Tissue Oxygen Saturation [StO2]. MI is able to detect the concentration of [Hb-total], [Hb-deoxy] & [Hb-O2] in absolute amounts in units of millimoles / unit volume of tissue measured. MI is also able to determine the percent fraction of mass, which is comprised of H2O in terms of percent mass.11, 14. This feature is critical to the performance of MI as a quantitative diagnostic method and, when combined with its tomographic capabilities, underscores the uniqueness of the method, and its potential use as a monitoring and diagnostic device to evaluate tissue transfer flaps after reconstructive surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients planned to undergo reconstructive surgery using either a pedicle or free tissue transfer flap seen by The Plastic Surgery Service on either an in-patient or outpatient bases.
* Adult patients that are planned to undergo reconstructive surgery as above and able to receive information regarding the study and provide informed consent to enrollment in the study.

Exclusion Criteria

* All emergency reconstructive surgery patients.
* Patients planned to undergo radiation therapy in the region of the reconstructive surgery within 6 months after surgery.
* Patients who develop hypotension requiring the administration of vasopressors either intra-operatively or during the post-operative period prior to discharge from the hospital.
* Patients who develop clinical signs of a surgical site infection at the location of the tissue transfer flap(s).
* Patients with the development of post-operative anemia requiring a blood transfusion during the first 72 hours after surgery.
* Patients with tattooing or pigmented lesions on the tissue transfer flap.
* Patients who incur injury to the flaps secondary to trauma within 6 months of the reconstructive surgery; with trauma defined as either accidental major trauma resulting in injury to the tissue transfer flap or surgical trauma as a result of further oncologic resection of tissues in close proximity to the tissue transfer flap.
* Minor under the age of 18 years of age.
* Patients deemed unable to comprehend and provide informed consent to enrollment into study due to either a cognitive deficit or medical condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects will be recruited from the pool of the patients seen in the Aesthetic and Plastic Surgery Institute clinics, as well as patients initially seen as in-patient consultations by the Plastic Surgery Service. Patients requiring reconstructive surgery using either a pedicle or free tissue transfer flap(s) will be identified. Patients requiring emergency reconstructive surgery after acute trauma will be excluded from the study as a matter of patient safety. The location and type of tissue transfer flaps enrolled will be dependent on the patient mix that presents during the study enrolment period. After explaining the nature, rationale, objectives, benefits, and risks of the study to the patients, they will be asked to consent to the study.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
detection of flap complications by modulated imaging compared to clinical standards | as long as hospital stay (baseline before surgery, 72 hours after surgery and before discharge from hospital)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory RD Evans, MD, FACS, Principal Investigator — Aesthetic and Plastic Surgery Institute
Locations (2):
- United States (2):
  - Aesthetic and Plastic Surgery Institute, Orange, California
  - The University of California Irvine, Orange, California